CLINICAL TRIAL: NCT01478529
Title: A Single Dose, Open Label, Randomized, Two-period Cross Over Study in Healthy Male Subjects to Assess the Absolute Bioavailability of YM178 OCAS-M Formulation
Brief Title: A Study to Find Out How Much Mirabegron Gets Into the Body After Dosing With a Tablet Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 178-CL-033
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Pharmacokinetics of Mirabegron; Bioavailability; Healthy Subjects
Keywords: Pharmacokinetics; Mirabegron; Phase 1
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm A (Experimental): low dose of mirabegron
  Interventions: Drug: mirabegron OCAS; Drug: mirabegron
- Treatment Arm B (Experimental): high dose of mirabegron
  Interventions: Drug: mirabegron OCAS; Drug: mirabegron

INTERVENTIONS:
Drug: mirabegron OCAS — oral administration
  Other Names: YM178 OCAS
Drug: mirabegron — iv administration
  Other Names: YM178

SUMMARY:
A study to evaluate how much of the active compound of mirabegron comes into the blood circulation when given as a controlled-release pill as compared to given intravenously.

DETAILED DESCRIPTION:
All participants will receive both oral and iv formulations, separated by a washout period. Treatment arm A will receive a lower dose of mirabegron; Treatment arm B will receive a higher dose of mirabegron.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 60.0 and 100.0 kg and Body Mass Index between 18.0 and 30.0 kg/m2

Exclusion Criteria:

* Known or suspected hypersensitivity to β-adrenergic receptor agonists or constituents of the formulations used
* Clinically significant elevation of serum creatinine or liver enzymes as evidenced by creatinine >150 ųmol/L; ASAT, ALAT or LDH> 2x ULN; ɣ-GT > 3x ULN and/or abnormal serum bilirubin
* Any clinically significant history of asthma, eczema, any other allergic condition or previous severe hypersensitivity to any drug
* Subjects taking β blockers or β agonists (eye drops allowed)
* Any clinically significant history of upper gastrointestinal symptoms (such as nausea, vomiting, abdominal discomfort or upset, or heartburn) in the 4 weeks prior to the first admission to the Research Unit
* Any clinically significant history of any other disease or disorder - gastrointestinal, cardiovascular, respiratory, ophthalmologic, renal, hepatic, neurological, dermatological, psychiatric or metabolic
* Any clinically significant abnormality following the investigator's review of the pre-study physical examination, ECG and clinical laboratory tests
* QTcB interval of > 430 (mean QTcB of two measurements > 430msec)
* Abnormal pulse rate measurement (<40 or >90 bpm) at the pre-study visit after subject has been resting in supine position for 5 min.
* Abnormal blood pressure measurements taken at the pre-study visit after subject has been resting in supine position for 5 min as follows:

  * Systolic blood pressure <95 or >160 mmHg
  * Diastolic blood pressure <40 or >90 mmHg
* Positive orthostatic test at screening i.e. any symptoms of dizziness, light-headedness etc. and a fall of > 20 mmHg in systolic blood pressure after 2 min standing and an increase in pulse rate of ≥ 20 bpm
* Regular use of any prescribed or OTC drugs except paracetamol up to 3 g/day, in the 4 weeks prior to admission to the Research Unit OR any use of such drugs in the 2 weeks prior to first admission to the Research Unit

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-02; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetics of mirabegron assessed by plasma concentration | Pre-dose until 72 hours after dosing

SECONDARY OUTCOMES:
Monitoring of safety and tolerability through assessment of vital signs, Electrocardiogram (ECG), clinical safety laboratory and adverse events | Baseline until 72 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Pharma Bio Research, Zuidlaren, Netherlands

REFERENCES:
- [Background] Eltink C, Lee J, Schaddelee M, Zhang W, Kerbusch V, Meijer J, van Marle S, Grunenberg N, Kowalski D, Drogendijk T, Moy S, Iitsuka H, van Gelderen M, Matsushima H, Sawamoto T. Single dose pharmacokinetics and absolute bioavailability of mirabegron, a beta(3)-adrenoceptor agonist for treatment of overactive bladder. Int J Clin Pharmacol Ther. 2012 Nov;50(11):838-50. doi: 10.5414/CP201782. PMID 22943933